CLINICAL TRIAL: NCT05867862
Title: Implementation of a Program to Strengthen Oral Hygiene in Patient With Cleft Deformities : HBD-Fentes
Brief Title: Implementation of a Program to Strengthen Oral Hygiene in Patient With Cleft Deformities
Acronym: HBD-Fentes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC22_0683
Record Dates: First submitted 2023-01-23; First posted 2023-05-22 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Orofacial Cleft
Keywords: Cleft Lip with or without Cleft Palate; Oral hygiene

STUDY DESIGN:
Intervention Model Description: For the control group: the instructions regarding OH given to the children and their parents will be the same than the one usually given by the maxilla-facial surgeons or the orthodontists during their annual follow-up visits. If the patients are in need of dental care, they will be encouraged to contact their dentist.
  For the test group: a dental consultation of 30 to 45 minutes will be added to the annual visit with a dentist. During this consultation the children will be incited to have a better OH, oral and written explanations will be provided. The goal is to have the best understanding of the importance of a good OH and brushing technique from the children and the parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional dental care (No Intervention): The instructions regarding OH given to the children and their parents will be the same than the one usually given by the maxilla-facial surgeons or the orthodontists during their annual follow-up visits. If the patients are in need of dental care, they will be encouraged to contact their dentist.
- Oral hygiene improvement (Experimental): A dental consultation of 30 to 45 minutes will be added to the annual visit with a dentist. During this consultation the children will be incited to have a better OH, oral and written explanations will be provided. The goal is to have the best understanding of the importance of a good OH and brushing technique from the children and the parents.
  If dental treatments are needed, they will be done at the same time, or they will be programmed for another time at the center of dental care (CSD).
  Due to the fact that most patient live far away from Nantes and the hospital, teleconsultation for patient in the test groups will happen every 2 months, in order to try and keep the child and parent motivation to a maximum and also assess the OH of the patient.
  Interventions: Other: Test

INTERVENTIONS:
Other: Test — A dental consultation of 30 to 45 minutes will be added to the annual visit with a dentist.
  If dental treatments are needed, they will be done at the same time, or they will be programmed for another time at the center of dental care (CSD).
  Due to the fact that most patient live far away from Nantes and the hospital, teleconsultation for patient in the test groups will happen every 2 months
  Arms: Oral hygiene improvement

SUMMARY:
A thorough analysis of the literature shows that children with clefts have a lesser oral hygiene (OH) and dental health (DH) than children without facial malformations, which leads to an increased number of tooth decay on temporary and permanent tooth and a poor gingival health due to gingivitis or periodontitis. The incidence of tooth decay is corelated with the severity of the cleft, children with bilateral cleft lip (including the alveolar bone) have a higher rate of tooth decay. Despite the fact that carious lesions are decreasing in general population, its rate remain constant in children with cleft.

Children who suffer from cleft in the north-west region of France are treated within the center of competence of rare disorder in the Nantes's hospital (CCMR MAFACE); this center is a gathering of different professional health specialist (surgeon, speech specialist, gynecologist, orthodontists, pediatrician…) working together to maximize treatment for those patients from diagnosis (sometime antenatal) to adulthood.

The active file of patients treated for cleft in Nantes's CHU is quite important, allowing an easy recruitment.

The investigator would like to create a clinical study, assessing the impact implementing a special program to strengthen OH in patient with cleft whose follow-up is taking place in Nantes's CCMR MAFACE. It would be an epidemiologic, prospective, randomized, controlled, and monocentric study

DETAILED DESCRIPTION:
Clef are congenital defects of the oral sphere; there are different types of cleft : regarding the cleft of the primary palate, the investigator can find the cleft lip's that are either uni ou bi laterals and can affect the nostrils and /or the alveolar bone; the clefs of the secondary palate are velar clefs, clefts of the palate or both meaning they affect the hard palate and soft palate.

Clefts accounts for 1 in 800 birth (1). A thorough analysis of the literature shows that children with clefts have a lesser oral hygiene (OH) and dental health (DH) than children without facial malformations, which leads to an increased number of tooth decay on temporary and permanent tooth and a poor gingival health due to gingivitis or periodontitis. The incidence of tooth decay is corelated with the severity of the cleft, children with bilateral cleft lip (including the alveolar bone) have a higher rate of tooth decay. Despite the fact that carious lesions are decreasing in general population, its rate remain constant in children with cleft.

A systemic revue looking for solutions or special therapy that could exists in order to optimized the oral health and dental status of cleft patient, conclude that there is a real necessity to maximized their treatment but few studies focus on preventive strategies or the development of tools to make OH easier for those patients.

Children who suffer from cleft in the north-west region of France are treated within the center of competence of rare disorder in the Nantes's hospital (CCMR MAFACE); this center is a gathering of different professional health specialist (surgeon, speech specialist, gynecologist, orthodontists, pediatrician…) working together to maximize treatment for those patients from diagnosis (sometime antenatal) to adulthood.

The active file of patients treated for cleft in Nantes's CHU is quite important, allowing an easy recruitment.

The investigatoir would like to create a clinical study, assessing the impact implementing a special program to strengthen OH in patient with cleft whose follow-up is taking place in Nantes's CCMR MAFACE. It would be an epidemiologic, prospective, randomized, controlled, and monocentric study.

The main goal of this study is to assess the effects of the implementation of OH programs and regular dental follow-ups for children with clef and its effect on their OH status.

The primary criteria will be the evolution of the dental index, which is the DMF index (dmft/DMFT) There are numerous secondary objectives, that will result from the data driven analysis during the consultations, they will not lengthen the duration of the consultation and neither add extra interventions on the patient.

* Assess the contribution of the implementation of OH programs and regular dental follow-ups for children with clef and its effect on their gingival status.
* Assess the satisfaction of the dental care and the follow-ups by the patients and the parents.
* Assess the accessibility to dental care for children with cleft
* Assess the impact of familial eating and hygiene habits on OH and its evolution during the year of follow-up.
* Assess the influence of orthodontics appliance, syndromes and other conditions related to the cleft, malocclusion, bucco-nasal fistulas, dental anomalies, sweet medications and medication inducing hyposialie on tooth decay
* Assess preferential localization of tooth decay
* Assess the financial impact of this protocol

Children with a cleft lip and or palate uni ou bilateral, between the age of 3 and 15 years old, coming to the CCMR MAFACE for treatment will be offered the possibility to participate to this study.

If they accept, they will be randomly assigned to 2 different groups.

For the control group: the instructions regarding OH given to the children and their parents will be the same than the one usually given by the maxilla-facial surgeons or the orthodontists during their annual follow-up visits. If the patients are in need of dental care, they will be encouraged to contact their dentist.

For the test group: a consultation of 30 to 45 minutes will be added to the annual visit with a dentist. During this consultation the children will be incited to have a better OH, oral explanations will be provided as well as written ones. The goal is to have the best understanding of the importance of good OH and brushing technique from the children and the parents.

If dental treatments are needed, they will be done in the same time, or they will be programmed for another time at de the center of dental car of the hospital (CSD).

Patient in the test groups will also have tele-consultations every 2 months, in order to try and keep the child motivation to a maximum and also assess the OH of the patient, they will also have an extra consultation with the dentist at 6 months.

Regarding the primary objective, the 2 groups will have a carious record done at day 1, year 1 and year 2; the secondary objective will also be collected at those dates, and for the test groups extra data will be collected at 2 month, 4 month, 6 month, 8 month and 10 month.

The number of necessary subjects was calculated using two different studies using the same criteria of judgement, 54 patients are needed for this study, 27 in each group.

If the investigator can show a significant difference in the medical and dental care due to the implication of this program, the goal would be to generalize this course of treatment to all the children with cleft within the service of maxillar-surgery (CMF) in Nantes and then once it's a well-rounded system the investigators could implement this way of working nation wild.

On a local scale, this initiative and adding a regular dental consultation could allow the establishment of a day hospital for those patients, and therefore it would be more comfortable for the patients and the parents.

ELIGIBILITY:
Inclusion Criteria:

* Child between the age of 3 and 15 years of, affected with a cleft associated or not with other syndromes or disabilities, with a regular follow up in the service of maxilla-facial surgery
* Authorization to participate
* Possibility to have a translator if difficulties to communicate

Exclusion Criteria:

* Impossibility to understand information during more than one session
* Not in possession of social security
* Refusal to participate in the study

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
DMF index : Assess the effects of the implementation of OH programs and regular dental follow-ups for children with clef and its effect on their OH status. | 1 year
  The primary criteria of judgment is the evolution of the dental index, which is the DMF index (dmft/DMFT).
  The DMF index if the census of all decayed, missing of filled teeth for temporary and permanent teeth.

SECONDARY OUTCOMES:
Assess the contribution of the implementation of OH programs and regular dental follow-ups for children with clef and its effect on their gingival health using Silness and Loe index. | 1 year
  The gingival health will be analyzed thanks to the Silness and Loe index, using a specific type and number of teeth following the Ramjiford principle 16-21-24-36-41-44 and 55-51-64-75-71-84; if one element is missing than the contralateral teeth will be analyzed. The Silness and Loe index is collected thanks to a 17 or 6 probe at the junction between teeth and gum.
  0: absence of dental plaque
  1. thin layer of dental plaque, noticed only after probing
  2. moderate accumulation of dental plaque visible by the naked eye
  3. abundance of dental plaque.
  A high score means a bad outcome.
Assess the satisfaction of the dental care and the follow-ups received during this study by the patients and parents | 1 year
  The satisfaction of this new course of treatment will be evaluated independently for children and parents thanks to an adapted questionnaire given at the 1 year follow up consultation.
  On a score scale, a high score means a good outcome and satisfaction from the parent and the child
Assess the accessibility of dental care for children with cleft | 1 year
  Accessibility to dental care will be evaluated following Whether or not the child had a dental practitioner before the inclusion as YES and No answers
Assess the accessibility of dental care for children with cleft | 1 year
  Accessibility to dental care will be evaluated following Last appointment with a dentist using a scale in month, <6 month, > 6 month, >1 year
Assess the accessibility of dental care for children with cleft | 1 year
  Accessibility to dental care will be evaluated following Distance between the place of life and the nearest hospital or dentist able to treat the child using a scale in <50, 50-100 >100 km.
Assess the impact of this study of oral and food hygiene and its evolution during the year of follow-up. | 1 year
  The impact of this study on the food and oral hygiene will be done following 5 criteria:
  1. Novice eating habits during the study (snacking, excessive breast feeding…) using Yes or no answers
  2. Drinking of sweet and acids beverage using Yes or no answers
  3. Use of a manual or electric toothbrush using Yes or no answers
  4. Use of an appropriate toothpaste with the right amount of Fluor using Yes or no answers
  5. Toothbrushing made by a parent or the child using Yes or no answers
Assess the influence of orthodontics appliance on OH | 1 year
  The impact orthodontic appliances will allow us to create 2 groups: one with and one without that will be compared thanks to Gingival index using Silness and Loe index : a high score means bad outcome
Assess the influence of orthodontics appliance on OH | 1 year
  The impact orthodontic appliances will allow us to create 2 groups: one with and one without that will be compared thanks to Dental index using DMF index : a high score means bad outcome
Assess the influence on weather being a girl or a boy influence on the rigor of OH | 1 year
  Studding the influence of the sex will allow to create two groups girl Vs Boys and compared them thanks to
  1. Gingival index Using Silness and Loe index : a high score means bad outcome
  2. Dental index using DFM index : a high score means bad outcome
Assess the influence on weather being a girl or a boy influence on the rigor of OH | 1 year
  Studding the influence of the sex will allow to create two groups girl Vs Boys and compared them thanks to Gingival index Using Silness and Loe index : a high score means bad outcome
Assess the influence on weather being a girl or a boy influence on the rigor of OH | 1 year
  Studding the influence of the sex will allow to create two groups girl Vs Boys and compared them thanks to Dental index using DFM index : a high score means bad outcome
Assess preferential localization of tooth decay | 1 year
  The preferential localization of tooth decay will be studied thanks to
  a. Dental index
Assess the influence of syndromes and other conditions related to cleft malformation, or dental anomalies on OH | 1 year
  In order to assess the influence of syndromes, pathologies associated with cleft, handicap and dental anomalies, the population will be divides in different groups: on the one hand healthy VS syndrome and pathology, on the other hand dental abnormalities VS non abnormalities, and finally Handicap VS non handicaps. All the groups will be compared using the Gingival index using Silness and Loe index : a high score means bad outcome
Assess the influence of syndromes and other conditions related to cleft malformation, or dental anomalies on OH | 1 year
  In order to assess the influence of syndromes, pathologies associated with cleft, handicap and dental anomalies, the population will be divides in different groups: on the one hand healthy VS syndrome and pathology, on the other hand dental abnormalities VS non abnormalities, and finally Handicap VS non handicaps. All the groups will be compared using the Dental index using DFM index : a high score means bad outcome
Assess the impact of malocclusion on OH | 1 year
  The influence of malocclusion will be studied thanks to 2 groups, one with dento-maxillary abnormalities and one without compared thanks to Gingival index using Silness and Loe index : a high score means bad outcome
Assess the impact of malocclusion on OH | 1 year
  The influence of malocclusion will be studied thanks to 2 groups, one with dento-maxillary abnormalities and one without compared thanks to Dental index using DFM index : a high score means bad outcome
Assess the influence of residual bucco-nasal fistulas on OH | 1 year
  Remaining bucco-nasal fistulas will allow us to divide the patients in 2 groups and study them thanks to:
  Gingival index using Silness and Loe index : a high score means bad outcome
Assess the influence of residual bucco-nasal fistulas on OH | 1 year
  Remaining bucco-nasal fistulas will allow us to divide the patients in 2 groups and study them thanks to:
  Dental index using DFM index : a high score means bad outcome
Assess the influence of sweet medications and medication inducing hyposialie on tooth decay. | 1 year
  The impact of sweet and hyposialant treatment will be studied thanks to
  a. Dental index : a high score means bad outcome
Assess the effect of oral dysfunction on OH | 1 year
  In order to assess the impact of oral dysfunction, the investigator need to label patients with this dysfunction as soon as possible and therefore create 2 groups: With and without oral dysfunctions analyzed them thanks to :
  Gingival index using Silness and Loe index : a high score means bad outcome
Assess the effect of oral dysfunction on OH | 1 year
  In order to assess the impact of oral dysfunction, the investigator need to label patients with this dysfunction as soon as possible and therefore create 2 groups: With and without oral dysfunctions analyzed them thanks to :
  Dental index using DFM index : a high score means bad outcome
Assess the financial impact of this protocol | 1 year
  The financial cost of this study will be assessed thanks to the calculus of what would cost all the dental consultation and therapeutic acts.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boeffard C, Loin J, Clouet R, Gaudin A, Corre P, Prud'Homme T. Implementation of a program to strengthen oral hygiene in patient with cleft deformities: a prospective randomized controlled clinical trial. Trials. 2025 Jan 9;26(1):14. doi: 10.1186/s13063-024-08507-w. PMID 39789639